CLINICAL TRIAL: NCT06548737
Title: Clinical Outcomes Following Primary Intracerebral Hemorrhage：A Multicenter Cohort Study
Brief Title: Clinical Outcomes Following Primary Intracerebral Hemorrhage
Acronym: COPI
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The People's Hospital of Haiyan (Unknown); Taizhou First People's Hospital (Other); The First People's Hospital of Pinghu (Unknown); The 2nd People's Hospital of Quzhou (Unknown)
Responsible Party: Sponsor
Other Study IDs: ZJU
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-06

CONDITIONS: Stroke; Intracerebral Hemorrhage
Keywords: Primary intracerebral hemorrhage; Stroke; Outcomes
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with primary intracerebral hemorrhage: We included adult patients who (1) admitted for primary ICH; (2) underwent blood routine test (hemoglobin included) and CT scan as soon as they arrived at hospital; (3) were not treated with neurosurgical procedures. We excluded patients who (1) had ICH secondary to known causes, including trauma, intracranial neoplasm and systemic diseases, as well as anticoagulative agents; or had isolated intraventricular hemorrhage (IVH); (2) mRS >2 before the current ICH episode (according to past medical records or description from guardians.

SUMMARY:
The investigators design an observational multi-center cohort study to provide contemporary information on the prevalence, characteristics, risk stratification，cost-effective ,treatments and prognosis of Chinese hospitalized adult patients with primary intracerebral hemorrhage.

DETAILED DESCRIPTION:
This cohort was an analysis based on patients from six stroke centers: the 2nd Affiliated Hospital of Zhejiang University; the First People's Hospital of Pinghu, Jiaxing; the First People's Hospital of Taizhou; the People's Hospital of Haiyan, Jiaxing; Tiantai County People's Hospital, Taizhou; the 2nd People's Hospital of Quzhou (Please see more information of this cohort in supplement). All hospitals are located in Zhejiang Province. Patients' data were entered by local trained registrars using standardised protocols, and the overall process of case registration, monitoring of the data quality, and inquiry and correction of erroneous data was managed and supervised by a steering committee.

We included adult patients who (1) admitted for primary ICH ; (2) underwent blood routine test (hemoglobin included) and CT scan as soon as they arrived at hospital; (3) were not treated with neurosurgical procedures. We excluded patients who (1) had ICH secondary to known causes, including trauma, intracranial neoplasm and systemic diseases12, as well as anticoagulative agents; or had isolated intraventricular hemorrhage (IVH); (2) mRS >2 before the current ICH episode (according to past medical records or description from guardians.

This study was approved by human research ethic committees at all participating centers, and conducted in compliance with the principles set forward by the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

- We included adult patients who (1) admitted for primary ICH ; (2) underwent blood routine test (hemoglobin included) and CT scan as soon as they arrived at hospital; (3) were not treated with neurosurgical procedures.

Exclusion Criteria:

* We excluded patients who (1) had ICH secondary to known causes, including trauma, intracranial neoplasm and systemic diseases12, as well as anticoagulative agents; or had isolated intraventricular hemorrhage (IVH); (2) mRS >2 before the current ICH episode (according to past medical records or description from guardians.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute primary intracerebral hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2016-10-27 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause death | 5 years after ICH
  Patients die of any reasons
ICH recurrence | 5 years after ICH
  Patients had an another ICH after this ictus
3-month outcome | 3 months after ICH
  3-month outcome is measured using modified Rankin Scale (mRS) score

SECONDARY OUTCOMES:
hematoma volume | up to 5 hours (A few hours after ICH)
  The volume of hematoma according to CT scan at the baseline when patients arrived at the emergency room
hematoma expansion | within 48 hours after ICH
  Patients had another CT scan during 24-48 hours after the first CT, and hematoma volume growth exceeding 33% or absolute hematoma growth exceeding 6ml
cerebral small vessel diseases (CSVDs) | within 2 weeks after ICH
  cerebral small vessel diseases evaluated by MRI, including cortical superficial siderosis (cSS), white matter hyperintensity (WMH), cerebral microbleed (CMB), etc.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Gao, Dr, Study Chair — Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Jin YJ, Yu GS, Tang LL, Li JW, Lin Q, Wu J, Song ZJ, An HN, Ye XH, Liu CJ, Gao F, Tong LS. Sex-specific hemoglobin thresholds and longitudinal trajectories in intracerebral hemorrhage outcomes: a multicenter cohort study. BMC Neurol. 2025 Jul 10;25(1):287. doi: 10.1186/s12883-025-04254-w. PMID 40640707